CLINICAL TRIAL: NCT05838456
Title: Deep Learning Enabled Endovascular Stroke Therapy Screening in Community Hospitals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Sunil A. Sheth, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-MS-19-0630; UL1TR003167 (NIH)
Record Dates: First submitted 2023-04-17; First posted 2023-05-01 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Acute Ischemic Stroke (AIS)
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge cluster-randomized trial with 4 clusters (4 different hospitals). In a stepped wedge fashion over 3 month intervals, the 4 clusters will initiate use of the software package (Viz.AI). The order of implementation of the Viz.AI software at the four hospitals will be randomly determined.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Hospital 1 - 3 months with no Viz.AI software, then 12 months with Viz.AI software (Experimental)
  Interventions: Device: Viz.AI software
- Hospital 2 - 6 months with no Viz.AI software, then 9 months with Viz.AI software (Experimental)
  Interventions: Device: Viz.AI software
- Hospital 3 - 9 months with no Viz.AI software, then 6 months with Viz.AI software (Experimental)
  Interventions: Device: Viz.AI software
- Hospital 4 - 12 months with no Viz.AI software, then 3 months with Viz.AI software (Experimental)
  Interventions: Device: Viz.AI software

INTERVENTIONS:
Device: Viz.AI software — Viz.AI software performs artificial intelligence-based automated detection of large vessel occlusions and alerts the AIS care team.

SUMMARY:
After onset of Acute Ischemic Stroke (AIS), every minute of delay to treatment reduces the likelihood of a good clinical outcome. A key delay occurs in the time between completion of computed tomography (CT) angiography of the head and neck and interpretation in the setting of AIS care.

The purpose of this study is to assess the effect of incorporating Viz.AI software, which via via a machine-learning algorithm performs artificial intelligence-based automated detection of large vessel occlusions (LVO) on CT angiography (CTA) images and alerts the AIS care team (diagnosis and treatment decisions will be based on the clinical evaluation and review of the images by the treating physician, per routine standard of care). The hypothesis is that integration of the software into the AIS care pathway will reduce delays in treatment. A cluster-randomized stepped-wedge trial will be performed across 4 hospitals in the greater Houston area.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 18 years of age or older.
* Patients who present to the emergency department with signs and/or symptoms concerning for acute ischemic stroke.
* Patients who undergo CT angiography imaging
* Patients determined to have a large vessel occlusion acute ischemic stroke. This determination will be made based on official radiology report for the CT angiography imaging.

Exclusion Criteria:

* Patients with incomplete data on the electronic medical record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Sheth, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez-Gutierrez JC, Kim Y, Salazar-Marioni S, Tariq MB, Abdelkhaleq R, Niktabe A, Ballekere AN, Iyyangar AS, Le M, Azeem H, Miller CC, Tyson JE, Shaw S, Smith P, Cowan M, Gonzales I, McCullough LD, Barreto AD, Giancardo L, Sheth SA. Automated Large Vessel Occlusion Detection Software and Thrombectomy Treatment Times: A Cluster Randomized Clinical Trial. JAMA Neurol. 2023 Nov 1;80(11):1182-1190. doi: 10.1001/jamaneurol.2023.3206. PMID 37721738

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 443 were enrolled, but 200 were excluded before assignment to groups. This is a stepped wedge cluster-randomized trial with 4 clusters (4 different hospitals). In a stepped wedge fashion over 3 month intervals, the 4 clusters will initiate use of the software package (Viz.AI). Each participant was only part of the study for one single period, in other words, participants did not progress to future periods.
Units Other Than Participants: hospitals
Groups:
- Hospital 1 - 3 Months With no Viz.AI Software, Then 12 Months With Viz.AI Software: Hospital will have 3 months with no Viz.AI software then 12 months with Viz.AI software integrated into the care pathway. Viz.AI software performs artificial intelligence-based automated detection of large vessel occlusions on CT angiography (CTA) images and alerts the AIS care team.
- Hospital 2 - 6 Months With no Viz.AI Software, Then 9 Months With Viz.AI Software: Hospital will have 6 months with no Viz.AI software then 9 months with Viz.AI software integrated into the care pathway. Viz.AI software performs artificial intelligence-based automated detection of large vessel occlusions on CT angiography (CTA) images and alerts the AIS care team.
- Hospital 3 - 9 Months With no Viz.AI Software, Then 6 Months With Viz.AI Software: Hospital will have 9 months with no Viz.AI software then 6 months with Viz.AI software integrated into the care pathway. Viz.AI software performs artificial intelligence-based automated detection of large vessel occlusions on CT angiography (CTA) images and alerts the AIS care team.
- Hospital 4 - 12 Months With no Viz.AI Software, Then 3 Months With Viz.AI Software: Hospital will have 12 months with no Viz.AI software then 3 months with Viz.AI software integrated into the care pathway. Viz.AI software performs artificial intelligence-based automated detection of large vessel occlusions on CT angiography (CTA) images and alerts the AIS care team.
Period: Step 1: Months 1-3
Arm/Group | Hospital 1 - 3 Months With no Viz.AI Software, Then 12 Months With Viz.AI Software | Hospital 2 - 6 Months With no Viz.AI Software, Then 9 Months With Viz.AI Software | Hospital 3 - 9 Months With no Viz.AI Software, Then 6 Months With Viz.AI Software | Hospital 4 - 12 Months With no Viz.AI Software, Then 3 Months With Viz.AI Software
Started | 38; 1 hospitals | 8; 1 hospitals | 11; 1 hospitals | 23; 1 hospitals
Completed | 38; 1 hospitals | 8; 1 hospitals | 11; 1 hospitals | 23; 1 hospitals
Not Completed | 0; 0 hospitals | 0; 0 hospitals | 0; 0 hospitals | 0; 0 hospitals
Period: Step 2: Months 4-6
Arm/Group | Hospital 1 - 3 Months With no Viz.AI Software, Then 12 Months With Viz.AI Software | Hospital 2 - 6 Months With no Viz.AI Software, Then 9 Months With Viz.AI Software | Hospital 3 - 9 Months With no Viz.AI Software, Then 6 Months With Viz.AI Software | Hospital 4 - 12 Months With no Viz.AI Software, Then 3 Months With Viz.AI Software
Started | 9; 1 hospitals | 3; 1 hospitals | 4; 1 hospitals | 20; 1 hospitals
Completed | 9; 1 hospitals | 3; 1 hospitals | 4; 1 hospitals | 20; 1 hospitals
Not Completed | 0; 0 hospitals | 0; 0 hospitals | 0; 0 hospitals | 0; 0 hospitals
Period: Step 3: Months 7-9
Arm/Group | Hospital 1 - 3 Months With no Viz.AI Software, Then 12 Months With Viz.AI Software | Hospital 2 - 6 Months With no Viz.AI Software, Then 9 Months With Viz.AI Software | Hospital 3 - 9 Months With no Viz.AI Software, Then 6 Months With Viz.AI Software | Hospital 4 - 12 Months With no Viz.AI Software, Then 3 Months With Viz.AI Software
Started | 11; 1 hospitals | 2; 1 hospitals | 5; 1 hospitals | 19; 1 hospitals
Completed | 11; 1 hospitals | 2; 1 hospitals | 5; 1 hospitals | 19; 1 hospitals
Not Completed | 0; 0 hospitals | 0; 0 hospitals | 0; 0 hospitals | 0; 0 hospitals
Period: Step 4: Months 10-12
Arm/Group | Hospital 1 - 3 Months With no Viz.AI Software, Then 12 Months With Viz.AI Software | Hospital 2 - 6 Months With no Viz.AI Software, Then 9 Months With Viz.AI Software | Hospital 3 - 9 Months With no Viz.AI Software, Then 6 Months With Viz.AI Software | Hospital 4 - 12 Months With no Viz.AI Software, Then 3 Months With Viz.AI Software
Started | 7; 1 hospitals | 2; 1 hospitals | 5; 1 hospitals | 9; 1 hospitals
Completed | 7; 1 hospitals | 2; 1 hospitals | 5; 1 hospitals | 9; 1 hospitals
Not Completed | 0; 0 hospitals | 0; 0 hospitals | 0; 0 hospitals | 0; 0 hospitals
Period: Step 4: Months 13-15
Arm/Group | Hospital 1 - 3 Months With no Viz.AI Software, Then 12 Months With Viz.AI Software | Hospital 2 - 6 Months With no Viz.AI Software, Then 9 Months With Viz.AI Software | Hospital 3 - 9 Months With no Viz.AI Software, Then 6 Months With Viz.AI Software | Hospital 4 - 12 Months With no Viz.AI Software, Then 3 Months With Viz.AI Software
Started | 16; 1 hospitals | 7; 1 hospitals | 10; 1 hospitals | 34; 1 hospitals
Completed | 16; 1 hospitals | 7; 1 hospitals | 10; 1 hospitals | 34; 1 hospitals
Not Completed | 0; 0 hospitals | 0; 0 hospitals | 0; 0 hospitals | 0; 0 hospitals

BASELINE CHARACTERISTICS:
Groups:
- no Viz.AI Software: Time before Viz.AI software was implemented
- With Viz.AI Software: Time after Viz.AI software was implemented. Viz.AI software performs artificial intelligence-based automated detection of large vessel occlusions and alerts the AIS care team.
- Total: Total of all reporting groups
Arm/Group | no Viz.AI Software | With Viz.AI Software | Total
Number analyzed (Participants) | 140 | 103 | 243
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69.5 [58.5 to 78] | 71 [57 to 79] | 70 [58 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 49 | 122
  Male | 67 | 54 | 121
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity: White | 58 | 50 | 108
  Race and Ethnicity: Black | 42 | 27 | 69
  Race and Ethnicity: Hispanic | 25 | 16 | 41
  Race and Ethnicity: Asian | 7 | 6 | 13
  Race and Ethnicity: Other | 8 | 4 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 140 | 103 | 243
Number of participants with prior stroke [Count of Participants; unit: Participants] | 24 | 19 | 43
Number of participants with prior transient ischemic attack (TIA) [Count of Participants; unit: Participants] | 11 | 5 | 16
Number of Participants with hypertension [Count of Participants; unit: Participants] | 107 | 75 | 182
Number of participants with hyperlipidemia [Count of Participants; unit: Participants] | 55 | 33 | 88
Number of participants with atrial fibrillation [Count of Participants; unit: Participants] | 41 | 30 | 71
Number of participants with diabetes [Count of Participants; unit: Participants] | 46 | 23 | 69
Number of participants with history of smoking [Count of Participants; unit: Participants] | 28 | 23 | 51
Number of participants with congestive heart failure [Count of Participants; unit: Participants] | 15 | 12 | 27
Time from last known well to time of hospital arrival [Median (Inter-Quartile Range); unit: minutes] — "Last known well" is the time prior to hospital arrival at which it was witnessed or reported that the patient was last known to be without the signs and symptoms of the current stroke or at his or her baseline state of health.
  minutes | 131.5 [61 to 472] | 147 [65 to 569] | 132 [61 to 498]
Score on the NIH Stroke Scale (NIHSS) [Median (Inter-Quartile Range); unit: score on a scale] — NIHSS indicates stroke severity. The score on NIHSS ranges from 0 to 42, with a higher score indicating greater stroke severity:
  Very Severe: >25 Severe: 15 - 24 Mild to Moderately Severe: 5 - 14 Mild: 1 - 5
  score on a scale | 17 [11 to 23] | 16 [11 to 21] | 17 [11 to 22]
Score on the Alberta stroke program early CT score (ASPECTS) [Median (Inter-Quartile Range); unit: score on a scale] — The Alberta stroke program early CT score (ASPECTS) is a 10-point quantitative topographic CT scan score used for stroke patients. Total score ranges from 0-10, with a lower score indicating a greater number of brain regions affected by stroke. An ASPECTS score less than or equal to 7 predicts a worse functional outcome at 3 months as well as symptomatic hemorrhage.
  score on a scale | 9 [7 to 10] | 10 [8 to 10] | 9 [7 to 10]
Number of participants who received intravenous tissue plasminogen activator (tPA) [Count of Participants; unit: Participants] | 63 | 48 | 111

OUTCOME MEASURES:

1. Primary Outcome: Time From Emergency Room Arrival to Initiation of Endovascular Stroke Therapy ("Door-to-groin" Time)
Time Frame: from the time of emergency room arrival to the time of initiation of endovascular stroke therapy (about 97 minutes)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | no Viz.AI Software | With Viz.AI Software
Number analyzed (Participants) | 140 | 103
minutes | 100 [81 to 116] | 88 [65 to 110]

2. Secondary Outcome: Number of Patients Who Received With Endovascular Stroke Therapy
Time Frame: at the time of initiation of endovascular stroke therapy
Measure: Count of Participants; unit: Participants
Arm/Group | no Viz.AI Software | With Viz.AI Software
Number analyzed (Participants) | 140 | 103
Participants | 140 | 103

3. Secondary Outcome: Number of Patients With Good Functional Outcome Defined as Modified Rankin Score (mRS) of 0-2
Description: The modified Rankin Scale (mRS) is used to assess the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scales ranges from 0-6, as follows: 0 = No symptoms; 1 = No significant disability. Able to carry out all usual activities, despite some symptoms; 2 = Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities; 3 = Moderate disability. Requires some help, but able to walk unassisted; 4 = Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted; 5 = Severe disability. Requires constant nursing care and attention, bedridden, incontinent; 6 = Dead.
Time Frame: 90 days
Population: mRS data were not collected for 50 in the no Viz.AI software arm and 79 in the with Viz.AI software arm.
Measure: Count of Participants; unit: Participants
Arm/Group | no Viz.AI Software | With Viz.AI Software
Number analyzed (Participants) | 90 | 24
Participants | 29 | 10

4. Secondary Outcome: Hospital Length of Stay
Description: The number of days of inpatient hospitalization.
Time Frame: From the time of admission to the hospital to the time of discharge (about 7 days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | no Viz.AI Software | With Viz.AI Software
Number analyzed (Participants) | 140 | 103
days | 7 [4 to 12] | 6 [3 to 10]

5. Secondary Outcome: Number of Patients With Intracranial Hemorrhage (ICH)
Description: Number of participants with any intracranial hemorrhage (ICH) and symptomatic ICH (Defined by ECASS II criteria)
Time Frame: From the time of admission to the hospital to the time of discharge (about 7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | no Viz.AI Software | With Viz.AI Software
Number analyzed (Participants) | 140 | 103
Participants
  Non-Symptomatic ICH | 17 | 17
  Symptomatic ICH | 7 | 2

ADVERSE EVENTS:
Time Frame: From the time of admission to the hospital to the time of discharge (about 7 days)
Arm/Group | no Viz.AI Software | With Viz.AI Software
All-Cause Mortality (participants affected / at risk) | 44/140 | 13/103
Serious Adverse Events (participants affected / at risk) | 7/140 | 2/103
Other Adverse Events (participants affected / at risk) | 17/140 | 17/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | no Viz.AI Software (N=140) | With Viz.AI Software (N=103)
Symptomatic intracerebral hemorrhage (ICH) (Vascular disorders) | 7 (7) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | no Viz.AI Software (N=140) | With Viz.AI Software (N=103)
non-symptomatic intracerebral hemorrhage (ICH) (Vascular disorders) | 17 (17) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT05838456/Prot_000.pdf